CLINICAL TRIAL: NCT03103022
Title: Combination of Acetaminophen and Ibuprofen in the Management of Patent Ductus Arteriosus in Premature Infants: A Pilot Study
Brief Title: Combination of Acetaminophen and Ibuprofen in the Management of Patent Ductus Arteriosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601912 - Jax
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Patent Ductus Arteriosus; Neonate
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional Group (Experimental): Preterm infants who met the eligibility criteria will receive both oral acetaminophen and ibuprofen. Oral acetaminophen [160 mg/5ml concentration] will be administered every 6 hours with dose of 15 mg/kg/dose for a total of twelve doses and oral ibuprofen [100 mg/5 ml] at 10 mg/kg/dose on first day followed by 5 mg/kg/dose at 24 and 48 hours for a total of three doses
  Interventions: Drug: Acetaminophen; Drug: ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — Oral acetaminophen [160 mg/5ml concentration] will be administered every 6 hours with dose of 15 mg/kg/dose for a total of twelve doses
  Other Names: Tylenol
Drug: ibuprofen — Oral ibuprofen [100 mg/5 ml] at 10 mg/kg/dose on first day followed by 5 mg/kg/dose at 24 and 48 hours for a total of three doses
  Other Names: Motrin

SUMMARY:
Patent ductus arteriosus or PDA is a blood vessel that connects the right and left side of the heart that usually closes after birth but remains open in some premature infants born before 30 weeks' gestation. When this blood vessel remains open for a long time, it may cause problems such as bleeding in the lung and brain, lung injury due to prolonged need of ventilator, and poor kidney function. It sometimes becomes necessary to close this blood vessel in the preterm infant. Currently, this blood vessel can be closed either by medication or surgery. Pain medications such as Ibuprofen and Indomethacin are routinely used medications to close PDA. However, in the last 5 year, acetaminophen has been found as an alternative medication to close PDA in preterm infants. In multiple studies, acetaminophen is found to be a safe alternative medication with lower side effects than current standard management. Intravenous Ibuprofen is approved by FDA to treat PDA in preterm infants. Although not approved by FDA, oral ibuprofen is being used for the management of PDA. However, the success rate of a single medication is approximately 70%. Both medications have been used in the previous clinical studies to treat the same condition in the preterm infants and fewer side effects were reported. Mechanism of both medications to close PDA is different and may work more effectively together than single medication alone. In this study, the investigator are going to use these two medications (Ibuprofen and Acetaminophen) at the same time if the child needs treatment and is eligible to participate in this study. This study is based on the assumption that by using both medications at the same time, investigator can close this blood vessel more effectively than with either drug alone.

DETAILED DESCRIPTION:
The ductus arteriosus is an essential blood vessel that connects the pulmonary artery and the aorta in the fetus. The patent ductus arteriosus (PDA) allows oxygenated blood that returns from the placenta to bypass the lungs and supply the fetal systemic circulation. In fetal life, ductus remains open due to low partial pressure of oxygen, circulating or locally produced prostaglandins and local nitric oxide production. Constriction of ductal vascular smooth muscle (functional closure) occurs within few hours of delivery due to decrease level of prostaglandin and rising oxygen concentrations. Closure of ductus can be affected by several perinatal and postnatal factors such as growth restriction, sepsis, and fluid overload. Spontaneous PDA closure occurs in > 34% extreme premature infants compared to > 95% in infants with birth weight more than 1500 grams. In a prospective study, 65 infants less than 1500 g birth weight were closely followed by serial echocardiograms. Sensitivity of ductal tissue to oxygen and prostaglandin differs in preterm compared to term infants. Without sufficient physiologic hypoxia, the ductus may fail to close or may reopen after initial constriction. Several co-morbidities have been associated with prolonged patency of the ductus in preterm infants (e.g., prolonged ventilator support, bronchopulmonary dysplasia, pulmonary hemorrhage, impaired renal function, intraventricular hemorrhage and cerebral palsy). Preterm infants with uncomplicated respiratory course, PDA is commonly managed conservatively. Currently hemodynamically significant PDA are managed medically (indomethacin and ibuprofen) and surgically. Recently, acetaminophen has gained attention as an alternative for PDA management due to its low cost, wide availability and the potential for fewer side effects. In two randomized controlled trials comparing acetaminophen with ibuprofen, authors have shown comparable closure rate of PDA with acetaminophen.

To our knowledge, a combination of the drugs has not been used to treat PDA in preterm infants and prospective study has not been conducted or published to determine the effectiveness of a combination of ibuprofen and acetaminophen in the treatment of PDA. As both medications are metabolized through different organs (hepatic and renal), the investigator assume that incidence of adverse events should not be affected. The Investigator hypothesize that the combination of oral ibuprofen and oral acetaminophen will be more effective, because the mechanisms of action differ for the two medications and hence may produce therapeutic synergy.

ELIGIBILITY:
Inclusion Criteria:

1. Infant with gestational age 23 to 30 weeks at birth and birth weight between 500 - 1000 grams
2. Postnatal age less than equal to 14 days
3. Hemodynamically significant PDA as defined by any of the following:

   1. Increased ventilator support attributed by the clinician to be due to PDA
   2. Hypotension and/or widening pulse pressure requiring vasopressors
   3. Signs of congestive heart failure such as pulmonary congestion
4. Echocardiographic criteria:

   1. Ratio of the smallest ductal diameter to the ostium of the left pulmonary artery > 0.5

Exclusion Criteria:

1. PDA-dependent congenital heart disease
2. Prior treatment with prophylactic indomethacin
3. Significant hyperbilirubinemia requiring exchange transfusion
4. Active or suspected necrotizing enterocolitis (NEC) and/or intestinal perforation
5. Abnormal liver enzymes
6. Platelets count < 50000 /l and / or active intracranial or gastrointestinal bleeding or from any other site
7. Major congenital anomalies such as neural tube defect, chromosomal abnormality and gastrointestinal defect

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Ductal closing rate | within 24-48 hrs after completion of treatment.
  To determine the ductal closure rate on echocardiography after completion of a first treatment course.

SECONDARY OUTCOMES:
Rate of ductal reopening | From birth until discharge / 36 weeks post menstrual age
  Echocardiographic evidence of closure followed by later re-opening of ductus if further echocardiogram is indicated.
Neonatal outcomes - Sepsis | until discharge / 36 weeks post menstrual age
  late-onset sepsis duration of hospital stay and death. Late onset sepsis: Defined as clinical signs of sepsis associated with a positive blood culture after 3 days of age.
Neonatal outcomes - Necrotizing Enterocolitis | until discharge / 36 weeks post menstrual age
  Necrotizing Enterocolitis (NEC): defined as stage 2 or greater duration of hospital stay and death.
Neonatal outcomes - Bronchopulmonary Dysplasia | until discharge / 36 weeks post menstrual age
  Late-onset bronchopulmonary dysplasia (BPD) is defined as oxygen requirement at 36 weeks or discharge for less than 32 weeks gestational infants duration of hospital stay and death.
neonatal outcomes - Ventilator days | until discharge / 36 weeks post menstrual age
  The number of days that ventilator support is needed during hospitalization.
Neonatal outcomes- Intraventricular Hemorrhage | until discharge / 36 weeks post menstrual age
  Late-onset severe intraventricular hemorrhage (IVH): IVH grade 3 and 4 both duration of hospital stay and death.
Neonatal outcomes - Periventricular Leukomalacia | until discharge / 36 weeks post menstrual age
  late-onset periventricular leukomalacia information will be derived from routine head ultra sounds (US) at 36 weeks / discharge as a standard of care duration of hospital stay and death.
Neonatal outcomes - Retinopathy of Prematurity | until discharge / 36 weeks post menstrual age
  Retinopathy of prematurity (ROP): severity of ROP will be derived from eye examination by pediatric ophthalmologist duration of hospital stay and death
Nutritional status - Weight | until discharge / 36 weeks post menstrual age
  Weight in grams at birth and discharge or 36 weeks post menstrual age converted to percentile or Z score by using Fenton 2013 growth chart.
Nutritional status - Length | until discharge / 36 weeks post menstrual age
  length in centimeters (cm) at birth and discharge or 36 weeks post menstrual age converted to either percentile or Z score by using Fenton 2013 growth chart.
Nutritional status - Head Circumference | until discharge / 36 weeks post menstrual age
  Head circumference (HC) in cm at birth and discharge or 36 weeks post menstrual age converted to either percentile or Z score by using Fenton 2013 growth chart.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Wolfson Children's Hospital, Jacksonville, Florida
  - University of Florida, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prescott S, Keim-Malpass J. Patent Ductus Arteriosus in the Preterm Infant: Diagnostic and Treatment Options. Adv Neonatal Care. 2017 Feb;17(1):10-18. doi: 10.1097/ANC.0000000000000340. PMID 27740976
- [Background] Coceani F, Baragatti B. Mechanisms for ductus arteriosus closure. Semin Perinatol. 2012 Apr;36(2):92-7. doi: 10.1053/j.semperi.2011.09.018. PMID 22414879
- [Background] Koch J, Hensley G, Roy L, Brown S, Ramaciotti C, Rosenfeld CR. Prevalence of spontaneous closure of the ductus arteriosus in neonates at a birth weight of 1000 grams or less. Pediatrics. 2006 Apr;117(4):1113-21. doi: 10.1542/peds.2005-1528. PMID 16585305
- [Background] Nemerofsky SL, Parravicini E, Bateman D, Kleinman C, Polin RA, Lorenz JM. The ductus arteriosus rarely requires treatment in infants > 1000 grams. Am J Perinatol. 2008 Nov;25(10):661-6. doi: 10.1055/s-0028-1090594. Epub 2008 Oct 10. PMID 18850514
- [Background] Benitz WE. Treatment of persistent patent ductus arteriosus in preterm infants: time to accept the null hypothesis? J Perinatol. 2010 Apr;30(4):241-52. doi: 10.1038/jp.2010.3. Epub 2010 Feb 25. PMID 20182439
- [Background] Benitz WE; Committee on Fetus and Newborn, American Academy of Pediatrics. Patent Ductus Arteriosus in Preterm Infants. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-3730. Epub 2015 Dec 15. PMID 26672023
- [Background] Gokmen T, Erdeve O, Altug N, Oguz SS, Uras N, Dilmen U. Efficacy and safety of oral versus intravenous ibuprofen in very low birth weight preterm infants with patent ductus arteriosus. J Pediatr. 2011 Apr;158(4):549-554.e1. doi: 10.1016/j.jpeds.2010.10.008. Epub 2010 Nov 20. PMID 21094951
- [Background] Olgun H, Ceviz N, Kartal I, Caner I, Karacan M, Tastekin A, Becit N. Repeated Courses of Oral Ibuprofen in Premature Infants with Patent Ductus Arteriosus: Efficacy and Safety. Pediatr Neonatol. 2017 Feb;58(1):29-35. doi: 10.1016/j.pedneo.2015.04.017. Epub 2016 Apr 29. PMID 27238078
- [Background] Adamska E, Helwich E, Rutkowska M, Zacharska E, Piotrowska A. [Comparison of the efficacy of ibuprofen and indomethacin in the treatment of patent ductus arteriosus in prematurely born infants]. Med Wieku Rozwoj. 2005 Jul-Sep;9(3 Pt 1):335-54. Polish. PMID 16547381
- [Background] Erdeve O, Yurttutan S, Altug N, Ozdemir R, Gokmen T, Dilmen U, Oguz SS, Uras N. Oral versus intravenous ibuprofen for patent ductus arteriosus closure: a randomised controlled trial in extremely low birthweight infants. Arch Dis Child Fetal Neonatal Ed. 2012 Jul;97(4):F279-83. doi: 10.1136/archdischild-2011-300532. Epub 2011 Dec 5. PMID 22147286
- [Background] Ohlsson A, Shah SS. Ibuprofen for the prevention of patent ductus arteriosus in preterm and/or low birth weight infants. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD004213. doi: 10.1002/14651858.CD004213.pub3. PMID 21735396
- [Background] Neumann R, Schulzke SM, Buhrer C. Oral ibuprofen versus intravenous ibuprofen or intravenous indomethacin for the treatment of patent ductus arteriosus in preterm infants: a systematic review and meta-analysis. Neonatology. 2012;102(1):9-15. doi: 10.1159/000335332. Epub 2012 Mar 8. PMID 22414850
- [Background] Oncel MY, Yurttutan S, Uras N, Altug N, Ozdemir R, Ekmen S, Erdeve O, Dilmen U. An alternative drug (paracetamol) in the management of patent ductus arteriosus in ibuprofen-resistant or contraindicated preterm infants. Arch Dis Child Fetal Neonatal Ed. 2013 Jan;98(1):F94. doi: 10.1136/archdischild-2012-302044. Epub 2012 May 18. No abstract available. PMID 22611117
- [Background] Hammerman C, Bin-Nun A, Markovitch E, Schimmel MS, Kaplan M, Fink D. Ductal closure with paracetamol: a surprising new approach to patent ductus arteriosus treatment. Pediatrics. 2011 Dec;128(6):e1618-21. doi: 10.1542/peds.2011-0359. Epub 2011 Nov 7. PMID 22065264
- [Background] Yurttutan S, Oncel MY, Arayici S, Uras N, Altug N, Erdeve O, Dilmen U. A different first-choice drug in the medical management of patent ductus arteriosus: oral paracetamol. J Matern Fetal Neonatal Med. 2013 May;26(8):825-7. doi: 10.3109/14767058.2012.755162. Epub 2013 Jan 15. PMID 23205872
- [Background] Peterson RG. Consequences associated with nonnarcotic analgesics in the fetus and newborn. Fed Proc. 1985 Apr;44(7):2309-13. PMID 3884385
- [Background] Terrin G, Conte F, Scipione A, Bacchio E, Conti MG, Ferro R, Ventriglia F, De Curtis M. Efficacy of paracetamol for the treatment of patent ductus arteriosus in preterm neonates. Ital J Pediatr. 2014 Feb 20;40(1):21. doi: 10.1186/1824-7288-40-21. PMID 24555510
- [Background] Green K, Drvota V, Vesterqvist O. Pronounced reduction of in vivo prostacyclin synthesis in humans by acetaminophen (paracetamol). Prostaglandins. 1989 Mar;37(3):311-5. doi: 10.1016/0090-6980(89)90001-4. PMID 2664901
- [Background] Anderson BJ. Paracetamol (Acetaminophen): mechanisms of action. Paediatr Anaesth. 2008 Oct;18(10):915-21. doi: 10.1111/j.1460-9592.2008.02764.x. PMID 18811827
- [Background] Dang D, Wang D, Zhang C, Zhou W, Zhou Q, Wu H. Comparison of oral paracetamol versus ibuprofen in premature infants with patent ductus arteriosus: a randomized controlled trial. PLoS One. 2013 Nov 4;8(11):e77888. doi: 10.1371/journal.pone.0077888. eCollection 2013. PMID 24223740
- [Background] Oncel MY, Yurttutan S, Erdeve O, Uras N, Altug N, Oguz SS, Canpolat FE, Dilmen U. Oral paracetamol versus oral ibuprofen in the management of patent ductus arteriosus in preterm infants: a randomized controlled trial. J Pediatr. 2014 Mar;164(3):510-4.e1. doi: 10.1016/j.jpeds.2013.11.008. Epub 2013 Dec 18. PMID 24359938
- [Background] Le J, Gales MA, Gales BJ. Acetaminophen for patent ductus arteriosus. Ann Pharmacother. 2015 Feb;49(2):241-6. doi: 10.1177/1060028014557564. Epub 2014 Oct 28. PMID 25352038
- [Background] Tekgunduz KS, Ceviz N, Demirelli Y, Olgun H, Caner I, Sahin IO, Yolcu C. Intravenous paracetamol for patent ductus arteriosus in premature infants - a lower dose is also effective. Concerning the article by M.Y. Oncel et al: Intravenous paracetamol treatment in the management of patent ductus arteriosus in extremely low birth weight infants [Neonatology 2013;103:166-169]. Neonatology. 2013;104(1):6-7. doi: 10.1159/000348568. Epub 2013 Mar 26. No abstract available. PMID 23548678
- [Background] El-Mashad AE, El-Mahdy H, El Amrousy D, Elgendy M. Comparative study of the efficacy and safety of paracetamol, ibuprofen, and indomethacin in closure of patent ductus arteriosus in preterm neonates. Eur J Pediatr. 2017 Feb;176(2):233-240. doi: 10.1007/s00431-016-2830-7. Epub 2016 Dec 21. PMID 28004188
- [Background] Oncel MY, Erdeve O. Oral medications regarding their safety and efficacy in the management of patent ductus arteriosus. World J Clin Pediatr. 2016 Feb 8;5(1):75-81. doi: 10.5409/wjcp.v5.i1.75. eCollection 2016 Feb 8. PMID 26862505
- [Background] Romagnoli C, De Carolis MP, Papacci P, Polimeni V, Luciano R, Piersigilli F, Delogu AB, Tortorolo G. Effects of prophylactic ibuprofen on cerebral and renal hemodynamics in very preterm neonates. Clin Pharmacol Ther. 2000 Jun;67(6):676-83. doi: 10.1067/mcp.2000.107048. PMID 10872650
- [Background] Peng S, Duggan A. Gastrointestinal adverse effects of non-steroidal anti-inflammatory drugs. Expert Opin Drug Saf. 2005 Mar;4(2):157-69. doi: 10.1517/14740338.4.2.157. PMID 15794710
- [Background] Kessel I, Waisman D, Lavie-Nevo K, Golzman M, Lorber A, Rotschild A. Paracetamol effectiveness, safety and blood level monitoring during patent ductus arteriosus closure: a case series. J Matern Fetal Neonatal Med. 2014 Nov;27(16):1719-21. doi: 10.3109/14767058.2013.871630. Epub 2014 Feb 7. PMID 24460433
- [Background] Walsh MC, Kliegman RM. Necrotizing enterocolitis: treatment based on staging criteria. Pediatr Clin North Am. 1986 Feb;33(1):179-201. doi: 10.1016/s0031-3955(16)34975-6. PMID 3081865
- [Background] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Background] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190
- [Background] Ramos FG, Rosenfeld CR, Roy L, Koch J, Ramaciotti C. Echocardiographic predictors of symptomatic patent ductus arteriosus in extremely-low-birth-weight preterm neonates. J Perinatol. 2010 Aug;30(8):535-9. doi: 10.1038/jp.2010.14. Epub 2010 Feb 25. PMID 20182434